CLINICAL TRIAL: NCT01431417
Title: Validation of a Kinematic Functional Shoulder Score Including Only Essential Movements
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FNS-DORE 13DPD6_135061
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Rotator Cuff, Syndrome; Frozen Shoulder; Humerus, Fracture; Other Instability of Joint, Shoulder Region
Keywords: Shoulder; Outcome treatment; Validation Studies as topic; Biomechanics; Shoulder, Joint Instability
MeSH Terms: conditions — Syndrome; Bursitis; Humeral Fractures; Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy volunteers: Healthy volunteers, less than 35 years old and presenting with no shoulder condition
- Patients with rotator cuff condition: Patients with rotator cuff condition, conservative treatment indicated
- Patients with shoulder instability: Patients with shoulder instability, conservative treatment indicated
- Patients with proximal humerus fracture: Patients with diaphyseal humerus fracture or subcapital humerus fracture treated surgically or conservatively, at 6 weeks post stabilization. (Surgical and conservative treatment will be considered as the same population from the functional point of view as functional outcome is similar) (Handoll et al. 2003).
- Patients with frozen shoulder: Patients with frozen shoulder, conservative treatment indicated

SUMMARY:
A lot of shoulder function evaluation scores exist but none has been universally accepted as a gold standard.

Recent studies have demonstrated the potential of computerized movement analysis with embedded sensors for objective evaluation of shoulder functional outcome following surgery.

A very simple testing procedure is possible as just a few repetitions of two simple shoulder movements are sufficient. This could potentially facilitate implementation of shoulder function movement analysis in current clinical practice.

However, at the present stage of development, the method needs to be extensively validated. This means that the research will intend to determine precisely for which current shoulder pathology it can be applied, what the outcome of healthy people is, what the reliability of the score is and how it can monitor patient evolution.

DETAILED DESCRIPTION:
Measurement of shoulder function is a controversial issue. There is a great variety of measurement tools but none of them has been universally accepted. There is therefore a need to develop extensively validated and convenient measurement tools.

Embedded computerized movement analysis can potentially meet these requirements for measurement of shoulder function. Ambulatory measurement devices allow application in various clinical conditions, display adequate precision and accuracy, and are considerably more straightforward than laboratory-based systems.

Using a Physilog ® II embedded system, Coley (2007) developed a relatively simple score of shoulder function (P Score). The method is based on arm power measurement by three-dimensional accelerometers and gyroscopes during seven consecutive shoulder movements. It demonstrated reliability, responsiveness and criterion-based validity. However, additional knowledge and technological progress could now contribute to further simplification of the testing procedure.

Indeed, a secondary analysis of Coley's study data based on principal component analysis and multiple regressions highlighted that a procedure including only two selected movements produces comparable results to P Score. Moreover, the development of wireless systems considerably simplifies set up. Consequently, simpler but equivalent measurement procedure can now be considered.

A pilot study (ClinicalTrials.gov identifier: NCT01281085) has been conducted to prepare this study. it contributed to determine the number of replications of movements needed and to refine the testing procedure.

The aim of this study is to proceed to an extensive validation study of the simplified testing procedure. Kinematic measurements will be carried out with four groups of patients presenting with frequent shoulder conditions (rotator cuff condition, shoulder instability, diaphyseal or subcapital humerus fracture, frozen shoulder) and a group of healthy people. Measurement procedure includes two consecutive measurements, alternatively conducted by two evaluators and measured simultaneously by two different movement analysis systems. Currently used functional questionnaires will be completed at both stages for comparison. Measurement will be performed at baseline and 6 months later.

Statistical analysis will address reproducibility, responsiveness, minimal clinically important difference and correlation with current clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff condition, conservative treatment indicated
* Shoulder instability, conservative treatment indicated
* Diaphyseal humerus fracture or subcapital humerus fracture treated surgically or conservatively, at 6 weeks post stabilization. (Surgical and conservative treatment will be considered as the same population from the functional point of view as functional outcome is similar) (Handoll et al. 2003).
* Frozen shoulder, conservative treatment indicated

Exclusion Criteria:

* Bilateral shoulder condition or other shoulder condition than the ones mentioned in inclusion criteria
* Any concomitant pain or condition involving upper limb
* Cervical spine condition involving upper limb pain or mobility restriction
* Insufficient French language level to understand patient information form, consent form or questionnaires
* Insufficient ability to give truly informed consent or to understand questionnaires. It will be proceeded to a Mini Mental State score in case of uncertainty, with exclusion criteria at 24 points/30 (ANAES 2000).
* Medical contraindication to execute movements required for score completion
* Tumor
* Neurological condition interfering with test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients consulting at the specialized shoulder consultation of the University Hospital of Lausanne
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Kinematic functional score | Baseline
  The kinematic functional score will be determined as the percentage of power of the pathological shoulder compared to the healthy shoulder (e.g. 70% means that the power developed during the movement of the pathological shoulder reaches 70% of the power developed on the healthy side)
Changes in kinematic functional shoulder scores | Change from Baseline in kinematic functional shoulder scores at 6 months
  Aforementioned score will be measured again 6 months after baseline to evaluate its responsiveness to patients' evolution

SECONDARY OUTCOMES:
Functional scores as determined by several currently used shoulder scores | Baseline
  Questionnaires include Constant score, Quick DASH, subjective shoulder value, Simple shoulder test, WOSI (Western Ontario Shoulder Instability Index; when relevant i.e. for shoulder instability), stiffness and pain EVA
Changes in functional shoulder scores | Change from Baseline in functional shoulder scores at 6 months
  All aforementioned scores will be measured again 6 months after baseline to compare their respective responsiveness to patients' evolution

CONTACTS AND LOCATIONS:
Overall Officials: Claude A. Pichonnaz, PT MSc, Study Director — HESAV and University Hospital of Lausanne; Farron Alain, MER PD, Study Chair — University of Lausanne Hospitals
Locations (1):
- Département de l'Appareil Locomoteur - CHUV, Lausanne, Switzerland

REFERENCES:
- [Background] Coley B, Jolles BM, Farron A, Bourgeois A, Nussbaumer F, Pichonnaz C, Aminian K. Outcome evaluation in shoulder surgery using 3D kinematics sensors. Gait Posture. 2007 Apr;25(4):523-32. doi: 10.1016/j.gaitpost.2006.06.016. Epub 2006 Aug 28. PMID 16934979
- [Background] Jolles BM, Duc C, Coley B, Aminian K, Pichonnaz C, Bassin JP, Farron A. Objective evaluation of shoulder function using body-fixed sensors: a new way to detect early treatment failures? J Shoulder Elbow Surg. 2011 Oct;20(7):1074-81. doi: 10.1016/j.jse.2011.05.026. PMID 21925353
- See also: Lay summary in French language on the sponsor's website (Swiss National Science Foundation) — http://p3.snf.ch/project-135061